CLINICAL TRIAL: NCT06365489
Title: Comparison of Brachial Wrist Index Before and After Implantation of Arteriovenous Fistulas, Based on Brachial Artery in Surgical Candidates Referred to Surgical Clinics in Gorgan in 1400
Brief Title: Comparison of Brachial Wrist Index Before and After Implantation of Arteriovenous Fistulas, Based on Brachial Artery
Status: Completed | Type: Observational
Sponsor: Golestan University of Medical sciences (Other)
Responsible Party: Principal Investigator, Pezhman Kharazm, MD, Vascular Surgeon, Golestan University of Medical sciences
Other Study IDs: 113293
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Vascular Access Complication
Keywords: Hemodialysis; Arterio Venous Fistula; Steal Syndrome; Wrist-Brachial Index; Vascular Access
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Arterio-Venous Fistula (AVF) is the most recommended vascular access for hemodialysis. Steal syndrome is a potential complication of AVF implantation and occurs secondary to diversion of the arterial flow of a limb to the venous system resulting in limb ischemia. Measuring wrist pressure compared to arm pressure before and after fistula implantation can be a suitable tool in predicting the possibility of Steal syndrome. In this study, the ratio of wrist to arm pressure and its relationship with Steal syndrome symptoms before and after fistula implantation are investigated.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) affects the structure and function of the kidneys. Many of CKD patients are not suitable candidates for a kidney transplant, so relying on some type of dyalisis is unavoidable.

Hemodialysis is the most common type of Renal Replacement Therapy. The best vascular access for hemodialysis in patients with chronic renal failure is Arterio-venous fistula (AVF). One of the complications of arterio-venous fistula is Steal syndrome which is ischemia of the limb secondary to blood flow diversion from the arterial system to the venous system through AVF.

Non-invasive wrist blood pressure measurement before and after the fistula construction may accurately assess the risk of ischemia and Steal syndrome from a functional AVF. Wrist-brachial index as a reliable prognostic test could be done easily in time of fistula construction and if it is normal, it assures the surgeon that the distal circulation is sufficient.

Summary of the project implementation method: First, the demographic questionnaire is completed for patients who meet the criteria for entering the study. Then the wrist-brachial index of patients who are candidates for fistula implantation before and after the fistula implantation is measured. Two weeks and three months later (times of suture removal and fistula maturation assessment), the measurements are repeated and their correlations with steal syndrome symptoms are recorded.

The data will be analyzed in SPSS16 statistical software

ELIGIBILITY:
Inclusion Criteria:

* ESRD patient candidate for hemodialysis
* Eligible for AVF implantation
* Cardiac Ejection Fraction > 20%
* Age> 18 years
* Suitable brachial artery and superficial vein for AVF

Exclusion Criteria:

* Death
* Non-consent of the patient
* Failure to follow up
* Fistula failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All ESRD patients who are candidates for AVF implantation after arterial and venous mapping, cardiac evaluation, and informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2022-12-11 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Early post operative WBI changes following AVF implantation | one year
  Comparison of wrist-brachial index before and after implantation of AVF in the operating room
Two-week post operative WBI changes following AVF implantation | one year
  Comparison of wrist-brachial index before and two-week after implantation of AVF.
Three-month post operative WBI changes following AVF implantation | one year
  Comparison of wrist-brachial index before and three-month after implantation of AVF.

SECONDARY OUTCOMES:
Correlation between WBI changes following AVF implantation with age | one year
  Comparison of WBI changes following AVF implantation in age sub groups
Correlation between WBI changes following AVF implantation with sex | one year
  Comparison of WBI changes following AVF implantation in sex sub groups
Correlation between WBI changes following AVF implantation with co-morbidities | one year
  Comparison of WBI changes following AVF implantation in co-morbidity sub groups
Correlation between WBI changes following AVF implantation with steal syndrome | one year
  comparison of WBI changes following AVF implantation between patients experiencing steal syndrome symptoms and Asymptomatic participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Pezhman Kharazm, MD, Gorgan, Golestan Province, Iran